CLINICAL TRIAL: NCT06106412
Title: Efficacy of Oocyte Activation With Two Types of Ca2+ Ionophore: a Prospective Randomized Study.
Brief Title: Efficacy of Oocyte Activation With Two Types of Ca2+ Ionophore.
Acronym: Calcifer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2303-VLC-043-MD
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Infertility, Female
Keywords: Artificial oocyte activation; Fertilization Failure; Calcium ionophore; Ionomycin; Calcimycin; Fertilization rate
MeSH Terms: conditions — Infertility, Female | interventions — Calcimycin

STUDY DESIGN:
Intervention Model Description: Prospective ranzomized analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 IONOMYCIN SIGMA (Experimental): The oocytes obtained from the patients allocated to this group will be subdivided again in two groups Group 1a: Oocytes treated with SIGMA ionomycin (treatment). Group 1b: Oocytes that will not be treated with any activator (Control).
  Interventions: Drug: Ionomycin SIGMA
- GROUP 2 A23187 (Active Comparator): The oocytes obtained from the patients allocated to this group will be subdivided again in two groups Group 2a: Oocytes treated with A23187 (treatment). Group 2b: Oocytes that will not be treated with any activator (Control).
  Interventions: Drug: A23187

INTERVENTIONS:
Drug: Ionomycin SIGMA — Oocytes will be activated with Ionomycin SIGMA
  Arms: GROUP 1 IONOMYCIN SIGMA
Drug: A23187 — Oocytes will be activated with A23187
  Arms: GROUP 2 A23187

SUMMARY:
This study is a prospective ranzomized analysis including 372 human oocytes from 44 women. Half of the oocytes from the same patient will be randomly allocated to induce oocyte activation using two protocols: in protocol nº 1 we will use ionomycin (prepared solution), protocol nª2 A23187 (GM508 CultActive Gynemed) will be applied. Non treated oocytes will serve as control. Oocyte fertilization rates, embryo development and embryo quality will be analyzed. Obstetrics variables of offspring will be also followed and compared.

DETAILED DESCRIPTION:
Background: Oocyte non-activation (OAD) is the main cause of fertilization failure in intracytoplasmic sperm injection (ICSI) cycles. Oocyte activation involves a series of consecutive events that take place in the oocyte during fertilization, triggered by the action of sperm-specific phospholipase C zeta (PLCz) that causes an increase in the amount of free Ca2+. This increase, as well as its transient elevations in space and time, is species-specific. Defects in this pattern of Ca2+ release and oscillation are attributed to most cases of OAD. Several strategies have been described and applied to achieve artificial oocyte activation (AOA), which use mechanical, electrical, or chemical stimuli, among which the use of calcium ionophores such as ionomycin and A23187 (calcimycin) predominates. Documented fertilization and pregnancy rates appear to be improved in patients with previous low fertilization rates or total fertilization failures after using ICSI-AOA compared to conventional ICSI. However, the lack of well-designed studies, the heterogeneity of the population undergoing AOA, and the scarcity of results comparing different AOA protocols make it difficult to assess the clinical efficacy and safety of the technique.

Study question: In patients with prior fertilization failure or low fertilization rates (30% or less), does AOA improve reproductive outcomes compared to conventional ICSI in patients with prior fertilization failure? and if it does, which protocol is more efficient?

ELIGIBILITY:
Inclusion Criteria:

* Own oocyte patients who have had previous fertilization failure in previous cycles.
* Own oocyte patients with fertilization rate in previous cycles less than or equal to 30% of the microinjected oocytes.

Exclusion Criteria:

* Oocyte Recipient Patients
* Sperm bank sperm recipient patients
* Patients who after oocyte decumulation have less than 2 mature oocytes.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in the percetage of usable blastocyst per injeected oocyte | 1 YEAR
  To evaluate which AOA protocol with the use of two calcium (Ca2+) ionophores, ionomycin and A23187 (calcimycin), is better (improvement from 15% to 25%)

SECONDARY OUTCOMES:
Sequencing unfertilized oocytes and arrested embryos using RNAseq | 1 year
  To quantify sequenced oocytes and arrested embryos after using RNAseq
Quantification of PLCZ in sperm cells by flow | 1 year
  To quantify PLCZ in sperm

CONTACTS AND LOCATIONS:
Locations (1):
- Ivirma Valencia, Valencia, Spain